CLINICAL TRIAL: NCT04016090
Title: An Evaluation of Folic Acid to Improve Endothelial Sensitivity to Shear Stress in Post-menopausal Women.
Brief Title: An Evaluation of Folic Acid to Improve Endothelial Sensitivity to Shear Stress in Seniors
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Montreal Heart Institute (Other)
Responsible Party: Principal Investigator, Daniel Gagnon, Principal Investigator, Montreal Heart Institute
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: ICM-2019-2596
Record Dates: First submitted 2019-07-03; First posted 2019-07-11 (Actual); Last update posted 2024-12-12 (Actual); Status verified 2024-12

CONDITIONS: Healthy Aging; Aging; Menopause
Keywords: Postmenopausal women; Vascular health; Folic acid
MeSH Terms: interventions — Folic Acid

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Placebo treatment (Placebo Comparator): Participant will be asked to ingest a placebo capsule.
  Interventions: Other: Placebo
- Folic Acid (Experimental): Participant will be asked to ingest a capsule containing 5 mg of folic acid.
  Interventions: Dietary Supplement: Folic Acid

INTERVENTIONS:
Dietary Supplement: Folic Acid — Folic acid (5 mg)
  Arms: Folic Acid
Other: Placebo — Placebo capsule
  Arms: Placebo treatment

SUMMARY:
The purpose of this study is to evaluate if folic acid improves endothelial sensitivity to shear stress in post-menopausal women.

DETAILED DESCRIPTION:
Cardiovascular diseases (CVD) have remained the leading cause of death globally for the last 15 years. Considering that advancing age is the primary risk factor for CVD, an increasingly aging population is expected to result in unprecedented levels of CVD. It therefore remains crucial to develop effective prevention or treatment strategies to reduce the impending health and economic burden of CVD.

Exercise is arguably the best intervention for the prevention and/or treatment of CVD. A key adaptation underlying the cardiovascular benefits of exercise is to offset and reverse age-related reductions in vascular function. Studies have demonstrated, at least in men, that active older adults demonstrate preserved vascular function relative to their sedentary peers and that exercise training interventions improve vascular function in previously sedentary older adults. However, these studies have almost exclusively been performed in men. In contrast, the few studies performed in older women consistently demonstrate that active women do not demonstrate preserved vascular function relative to their sedentary peers and that exercise training interventions do not improve vascular function in previously sedentary women. This observation has been attributed to the loss of oestrogens that accompanies menopause. Although the mechanisms have not been fully elicited, it is possible that the loss of oestrogens desensitizes the endothelium to the physiological stimuli that result in improved vascular function with exercise training. Indeed, exercise improves vascular function in previously sedentary older women when it is combined with oestrogen replacement. Nevertheless, chronic oestrogen replacement therapy is not a viable intervention as it is associated with an increased risk of breast cancer. Alternative solutions to restore the beneficial effects of exercise on vascular function in post-menopausal women are thus urgently needed.

The overall objective of this project is to determine if folic acid, an over-the-counter supplement that has been shown to provide beneficial vascular adaptations, can be used to improve vascular function in post-menopausal women. It is hypothesized that folic acid will improve blood vessel function in post-menopausal women and age-matched males.

ELIGIBILITY:
Inclusion Criteria:

* ≥ 1-year amenorrhea
* Body mass index ≤ 30 kg/m2
* Resting blood pressure < 140 / < 90 mmHg
* Non-smoker (≥ 1-year)

Exclusion Criteria:

* Diagnosis of cardiac, vascular, respiratory, neurological or metabolic disease and/or a prescription of medications for the treatment of such diseases.
* For female participants, hormonal replacement therapy within 1 year of enrolment in the study.
* For female participants, having undergone an ovariectomy.

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2019-09-09 (Actual); Primary Completion 2024-04-03 (Actual); Study Completion 2024-04-03 (Actual)

PRIMARY OUTCOMES:
Endothelial sensitivity to shear rate | Measured 2 hours after placebo or folic acid consumption
  Change in brachial artery diameter for given levels of shear rate during rhythmic handgrip exercise

SECONDARY OUTCOMES:
Neurovascular transduction | Measured 2 hours after placebo or folic acid consumption
  Change in femoral artery diameter for a given increase in muscle sympathetic nerve activity during isometric handgrip exercise to fatigue.

CONTACTS AND LOCATIONS:
Locations (1):
- Cardiovascular Prevention and Rehabilitation Centre of the Montreal Heart Institute, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No
All individual data will be de-identified and available to the public through publications, media articles and conference presentations